CLINICAL TRIAL: NCT00234533
Title: Phase IIIB, International, Single Group, Open Study to Define an Optimal Monitoring of IGF-1 in Children Treated With NutropinAq, Using a Novel Capillary Blood Collection Method
Brief Title: Study to Define Optimal IGF-1 Monitoring in Children Treated With NutropinAq
Acronym: OPTIMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-79-58035-700; 2004-000356-17 (EudraCT Number)
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Results first posted 2018-08-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Turner Syndrome; Renal Insufficiency, Chronic; Pituitary Diseases; Dwarfism
Keywords: growth; child development; growth hormone; inadequate growth hormone secretion; growth failure
MeSH Terms: conditions — Turner Syndrome; Renal Insufficiency, Chronic; Pituitary Diseases; Dwarfism; Failure to Thrive | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NutropinAq 10 mg/2 mL (30 IU) (Experimental): Patients received daily subcutaneous (s.c.) injections of NutropinAq 10 milligrams (mg)/2 milliliters (mL) for 6 months. The therapeutic daily doses administered were as follows:
  * GHD patients: 0.025 - 0.035 mg/ kilogram (kg) bodyweight
  * TS patients: up to 0.05 mg/kg bodyweight
  * CRI patients: up to 0.05 mg/kg bodyweight
  Patients visited the study clinic for a baseline visit and for 2 other visits every 3 months (Weeks 12 and 24). Additional home assessments were made at Weeks 21, 22 and 23.
  The investigator determined the dose administered to each patient, and it was recommended to perform the injection in the evening.
  Interventions: Drug: Somatropin (rDNA origin)

INTERVENTIONS:
Drug: Somatropin (rDNA origin) — Daily subcutaneous injections, 0,025 - 0,05 mg/kg/day for 6 months.

SUMMARY:
The main purpose of this study is to establish an optimal monitoring regimen in NutropinAq treated children, using newly developed capillary blood spot IGF-1 measurement technology.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 with growth failure associated with inadequate growth hormone secretion, or Turner syndrome or chronic renal insufficiency.

Exclusion Criteria:

* Children with closed epiphyses
* Children with active neoplasm
* Children with acute critical illness

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 251 (Actual)
Dates: Start 2004-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (45):
- Belgium (2):
  - Dienst Kindergeneeskunde, Brussels
  - Dienst Kindergeneeskunde, Edegem
- Klinika Deti a Dorostu, Prague, Czechia
- Denmark (2):
  - Aalborg Sygehus Nord, Borneafdelingen, Aalborg
  - Sygeh. i Ringkjobing Amt, Borneafdeling, Herning
- Helsinki University Central Hospital, Helsinki, Finland
- France (15):
  - CHU - Hôtel Dieu, Angers
  - Cabinet Médical, Bordeaux
  - CHU Grenoble, Grenoble
  - Centre Hospitalier General, Le Havre
  - CHU Timone Enfants, Marseille
  - CHU de Montpellier, Montpellier
  - Hôpital Archet 2, Nice
  - Hôpital Saint-Vincent de Paul, Paris
  - Groupe Hospitalier de Necker, Paris
  - Hôpital Charles Nicolle, Rouen
  - CHU Hautepierre, Strasbourg
  - Centre Hospitalier de Bigorre, Tarbes
  - Cabinet Médical, Toulouse
  - Hôpital des Enfants, Toulouse
  - Centre Pédiatrique Gatien de Clocheville, Tours
- Germany (2):
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Universitätsklinikum Tübingen, Tübingen
- Greece (2):
  - General State Hospital of Nikaia, Athens
  - PA Kyriakou Children's Hospital, Athens
- Italy (7):
  - Azienda Policlinico - Università di Catania, Catania
  - Ospedale Policlinico, Chieti
  - Clinica Pediatrica II, Florence
  - Il Università degli Studi di Napoli, Napoli
  - Clinica Pediatrica, Universita Federico II di Napoli, Napoli
  - Clinica Pediatrica, Novara
  - Clinica Pediatrica, Parma
- Institutul de Endocrinologie C.I. Parhon, Bucharest, Romania
- Russia (2):
  - Endocrinology Research Centre RAMS, Institute of Pediatric Endocrinology, Moscow
  - Tushino Pediatric Hospital, RMAPE Department of Endocrinology for Childhood and Adolescent Age, Moscow
- Il Detska Klinika, Bratislava, Slovakia
- Spain (5):
  - Hospital de Nens de Barcelona, Barcelona
  - Hospital General Universitario, Elche
  - Hospital Gregorio Marañón, Madrid
  - Hospital Parc Taulí, Sabadell
  - Hospital Clínico Universitario, Santiago de Compostela
- Ukraine (2):
  - Scientific-Research Institute of Endocrinology, Academy of Medical Science of Ukraine, Kiev
  - Ukrainian Scientific practical Centre of Endocrine surgery, Endocrine Organs and Tissues Transplantation, Kiev
- United Kingdom (2):
  - St George's Hospital, London, England
  - University Hospital Wales, Cardiff, Wales

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 251 children presenting growth failure associated with Growth Hormone Deficiency (GHD), Turner Syndrome (TS) or Chronic Renal Insufficiency (CRI) were screened (with informed consent) in 46 study centers across Europe. First patient enrolled: 7 June 2004; last subject completed: 22 July 2008
Pre-assignment Details: Of the 251 children screened 3 did not receive study medication, 1 due to withdrawal of consent, 1 did not meet screening criteria for height and 1 was not included due to the investigator's decision.
Groups:
- NutropinAq 10 mg/2 ml (30 IU): Patients received daily subcutaneous (s.c.) injections of NutropinAq 10 milligrams (mg)/ 2 milliliters (mL) for 6 months. The therapeutic daily doses administered were as follows:
  * GHD patients: 0.025 - 0.035 mg/ kilogram (kg) bodyweight
  * TS patients: up to 0.05 mg/kg bodyweight
  * CRI patients: up to 0.05 mg/kg bodyweight
  Patients visited the study clinic for a baseline visit and for 2 other visits every 3 months (Weeks 12 and 24). Additional home assessments were made at Weeks 21, 22 and 23.
  The investigator determined the dose administered to each patient, and it was recommended to perform the injection in the evening.
Period: Overall Study
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Started | 251
Completed | 240
Not Completed | 11
Not completed — Withdrawal by Subject | 6
Not completed — Adverse Event | 2
Not completed — Enrolled but not treated | 3

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) Population consisted of all treated patients (enrolled patients who received at least one injection of treatment) and who provided any follow-up data.
Groups:
- NutropinAq 10 mg/2 ml (30 IU): Patients received daily s.c. injections of NutropinAq 10 mg/ 2 mL for 6 months. The therapeutic daily doses administered were as follows:
  * GHD patients: 0.025 - 0.035 mg/kg bodyweight
  * TS patients: up to 0.05 mg/kg bodyweight
  * CRI patients: up to 0.05 mg/kg bodyweight
  Patients visited the study clinic for a baseline visit and for 2 other visits every 3 months (Weeks 12 and 24). Additional home assessments were made at Weeks 21, 22 and 23.
  The investigator determined the dose administered to each patient, and it was recommended to perform the injection in the evening.
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 106
Birth height [Mean (Standard Deviation); unit: centimeters (cm)] | 48.49 (3.36)
Birth weight [Mean (Standard Deviation); unit: kg] | 2.94 (0.60)
Duration of gestation [Mean (Standard Deviation); unit: weeks of amenorrhea] | 38.7 (2.6)
Genetic target height [Mean (Standard Deviation); unit: cm] — The genetic potential height, or target height was estimated using the adult height of each parent (i.e. genetic mother and father).
  cm | 166.26 (8.16)
Calculated genetic target height Standard Deviation Score (SDS) [Mean (Standard Deviation); unit: Standard Deviations (SD)] — The genetic potential height, or target height was estimated as follows:
  * Boys Target Height = [(mother height cm + father height cm)/2] + 6.5 cm.
  * Girls Target Height = [(mother height cm + father height cm)/2] - 6.5 cm. The French growth charts were used for the calculation of standard deviation score (SDS) parameters: the charts provide for each age range and sex a mean parameter and standard deviation (SD) value, from which the SDS parameter can be derived assuming a normal distribution. For example: Height SDS = (height - reference mean height (age, sex)) / reference SD (age, sex).
  Standard Deviations (SD) | -0.33 (0.95)
Duration of previous Growth Hormone (GH) treatment [Mean (Standard Deviation); unit: years] — Population: Data is presented for non-naïve patients only.
  years
    number analyzed (Participants) | 59
    (all) | 1.68 (1.56)
Auxological Parameter - Height [Mean (Standard Deviation); unit: cm] | 122.95 (20.24)
Auxological Parameter - Calculated height SDS [Mean (Standard Deviation); unit: SD] | -2.68 (1.33)
Auxological Parameter - Weight [Mean (Standard Deviation); unit: kg] | 27.97 (11.91)
Auxological Parameter - Calculated weight SDS [Mean (Standard Deviation); unit: SD] | -1.85 (1.88)
Auxological Parameter - Annualised Growth Velocity (GV) [Mean (Standard Deviation); unit: cm/year] | 4.94 (2.56)
Auxological Parameter - Calculated annualised GV SDS [Mean (Standard Deviation); unit: SD] | -0.56 (2.67)

OUTCOME MEASURES:

1. Primary Outcome: Insulin-Like Growth Factor I (IGF-I) Levels Measured Using the Timed Capillary Blood Spot Samples
Description: Fingertip capillary blood was collected using filter paper cards for the assay of capillary blood spot IGF-I in line with the monitoring recommendations of the Lawson Wilkins Paediatric Endocrine Society (LWPES) for treatment with recombinant GH therapy in children.
  Capillary IGF-I assays were performed by the patient at home one day per week during Weeks 21, 22 and 23 only (same week day). The samples were scheduled in the evening prior to the injection of NutropinAq and between 7:00 and 9:00 the following morning. An extended window from 6:00 to 12:00 was allowed for defining protocol deviations.
  The number of capillary blood spot IGF-I measurements and the optimal timing of samples to assess the IGF-I status of NutropinAq treated patients was assessed. IGF-I measurements for the morning and evening sampling are presented.
Time Frame: At Weeks 21, 22 and 23
Population: The ITT Population consisted of all treated patients (enrolled patients who received at least one injection of treatment) and who provided any follow-up data. Only evaluable subjects with an assessment at the specified timepoint were included in each individual analysis.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Groups:
- NutropinAq 10 mg/2 ml (30 IU): Patients received daily s.c. injections of NutropinAq 10 mg/ 2 mL for 6 months. The therapeutic daily doses administered were as follows:
  * GHD patients: 0.025 - 0.035 mg/ kilogram kg bodyweight
  * TS patients: up to 0.05 mg/kg bodyweight
  * CRI patients: up to 0.05 mg/kg bodyweight
  Patients visited the study clinic for a baseline visit and for 2 other visits every 3 months (Weeks 12 and 24). Additional home assessments were made at Weeks 21, 22 and 23.
  The investigator determined the dose administered to each patient, and it was recommended to perform the injection in the evening.
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
nanograms/milliliter (ng/mL)
  Week 21 Morning sampling: number analyzed (Participants) | 226
  Week 21 Morning sampling | 223.54 (161.86)
  Week 21 Evening sampling: number analyzed (Participants) | 230
  Week 21 Evening sampling | 212.97 (153.61)
  Week 22 Morning sampling: number analyzed (Participants) | 223
  Week 22 Morning sampling | 238.02 (177.89)
  Week 22 Evening sampling: number analyzed (Participants) | 229
  Week 22 Evening sampling | 226.90 (164.38)
  Week 23 Morning sampling: number analyzed (Participants) | 226
  Week 23 Morning sampling | 241.58 (167.75)
  Week 23 Evening sampling: number analyzed (Participants) | 225
  Week 23 Evening sampling | 235.47 (168.48)
Statistical Analysis 1: Comparison: NutropinAq 10 mg/2 ml (30 IU); An Intra-class Correlation Coefficient (ICC) for the evening series (defined as 12:00 to 24:00) was determined for the overall ITT population to confirm whether only one measurement would be sufficient to accurately represent the IGF-I measurement over Weeks 21, 22 and 23. The ICC expresses the relative magnitude of the 2 components of the total variability, i.e. the biological variability and random error, in a series of measurements on different patients; Test type: Other — An one-way Analysis of Covariance (ANOVA) was used to calculate the between patient variation and within patient variation and then the ICC and its confidence limitations; ICC = 0.90, 95% CI 2-sided [0.88 to 0.92] — An ICC ≥ 0.8 was considered satisfactory and indicative that a single sample would be representative of the overall IGF-I status
Statistical Analysis 2: Comparison: NutropinAq 10 mg/2 ml (30 IU); An ICC for the morning series (defined as 06:00 to 12:00) was determined for the overall ITT population to confirm whether only one measurement would be sufficient to accurately represent the IGF-I measurement over Weeks 21, 22 and 23. The ICC expresses the relative magnitude of the 2 components of the total variability, i.e. the biological variability and random error, in a series of measurements on different patients; Test type: Other — An one-way ANOVA was used to calculate the between patient variation and within patient variation and then the ICC and its confidence limitations; ICC = 0.92, 95% CI 2-sided [0.90 to 0.93] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Assessment of IGF-I Levels: Categorised by Weekly Timing (Weeks 21-23) and Daily Timing (Morning and Evening)
Description: The influence of daily and weekly timing on the IGF-I value as measured using the capillary blood spot method was analysed. A 3-way analyses of variance (ANOVA) was performed with patient, day and daily timing as factors after appropriate transformation to obtain normally distributed parameters. The interaction day*time was tested and kept in the model only if p-value<0.1. Parameter estimates from the statistical model are presented as least squares means for the categories of daily timing (Morning and Evening) and weekly timing (Week 21, Week 22 and Week 23). The values reported for Week 21, 22, and 23 represent the average IGF-I levels from the morning and evening samples at each week. The values reported for Evening represent the Evening IGF-I levels averaged across Weeks 21, 22, and 23, and similarly for the Morning values.
Time Frame: At Weeks 21, 22 and 23
Population: The ITT Population consisted of all treated patients (enrolled patients who received at least one injection of treatment) and who provided any follow-up data.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
ng/mL
  Week 21 | 218.3 [203.0 to 233.5]
  Week 22 | 232.4 [217.1 to 247.8]
  Week 23 | 238.5 [223.2 to 253.9]
  Evening | 225.1 [212.6 to 237.6]
  Morning | 234.4 [221.8 to 246.9]
Statistical Analysis 1: Comparison: NutropinAq 10 mg/2 ml (30 IU); Analysis of the weekly timing effect (Week 21 versus Week 22 versus Week 23) on the IGF-I value as measured by capillary blood spot method; Test type: Other; Fisher's F statistic (F) value = 1.79; For the effect of the weekly timing on the IGF-I levels; F value = 1.79 and the significance probability value, PR>F = 0.1678
Statistical Analysis 2: Comparison: NutropinAq 10 mg/2 ml (30 IU); Analysis of the daily timing effect (morning versus evening) on the IGF-I value as measured by capillary blood spot method; Test type: Other; F value = 1.06; For the effect of the daily timing on the IGF-I levels; F value = 1.06 and the significance probability value, PR>F = 0.3035

3. Secondary Outcome: Assessment of IGF-I Levels: Categorised by Sex and Prepubertal Status
Description: The influence of sex and prepubertal status on the IGF-I value as measured using the capillary blood spot method was analysed. Parameter estimates from the statistical model are presented as least squares means for the categories of sex (male and female) and prepubertal status (pubertal and prepubertal). The values reported represent average IGF-I levels as determined from the 6 measurements taken (i.e. morning and evening samples at Weeks 21, 22 and 23).
Time Frame: At Weeks 21, 22 and 23
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
ng/mL
  Female: number analyzed (Participants) | 138
  Female | 234.4 [224.7 to 244.4]
  Male: number analyzed (Participants) | 106
  Male | 172.1 [162.7 to 181.9]
  Pubertal: number analyzed (Participants) | 116
  Pubertal | 238.9 [224.8 to 253.5]
  Prepubertal: number analyzed (Participants) | 128
  Prepubertal | 168.4 [160.7 to 176.3]
Statistical Analysis 1: Comparison: NutropinAq 10 mg/2 ml (30 IU); Analysis of the effect of the patient's sex (male versus female) on the IGF-I value as measured by capillary blood spot method; Test type: Other; F value = 83.97; For the effect of the patient's sex on the IGF-I levels; F value = 83.97 and the significance probability value, PR>F = <0.0001
Statistical Analysis 2: Comparison: NutropinAq 10 mg/2 ml (30 IU); Analysis of the effect of the patient's pubertal status (pubertal versus prepubertal) on the IGF-I value as measured by capillary blood spot method; Test type: Other; F value = 68.35; For the effect of the patient's pubertal status on the IGF-I levels; F value = 68.35 and the significance probability value, PR>F = <0.0001

4. Secondary Outcome: Multivariate Linear Regression Analyses to Assess Factors Affecting the Variability of IGF-I Levels: Categorised by Disease Condition and Location
Description: A multivariate linear regression analysis of factors on within-subject coefficient of variation (WCV) using a stepwise forward-backward elimination was used to determine the effect of individual factors on IGF-I values as measured using the capillary blood spot method (p=0.15 for a variable to enter and remain in the model). The WCV was computed from the series of 6 measurements (2 samplings in each of Weeks 21, 22 and 23). The influence of disease condition and country clusters on the IGF-I value were assessed.
  Country clusters: cluster 1: France; cluster 2: Spain, Greece, Romania and Italy; cluster 3: UK, Belgium, Czech Republic, Denmark, Germany, Slovakia, Austria and Finland ; cluster 4: Russia ; cluster 5: Ukraine.
  Parameter estimates from the statistical model presented as least squares means for categories of disease condition (GHD and TS) and location (Clusters 1, 2, 3, 4 and 5) are presented.
Time Frame: Up to Week 24
Population: The ITT Population consisted of all treated patients (enrolled patients who received at least one injection of treatment) and who provided any follow-up data. Only evaluable subjects within each of the individual subgroups are presented for each category. As there was only 1 patient with CRI, no analysis was performed for this disease condition.
Measure: Least Squares Mean (Standard Error); unit: Regression coefficient
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
Regression coefficient
  Disease condition: GHD: number analyzed (Participants) | 158
  Disease condition: GHD | 0.058 (0.031)
  Disease condition: TS: number analyzed (Participants) | 85
  Disease condition: TS | 0.000 (0)
  Cluster 1: number analyzed (Participants) | 81
  Cluster 1 | 0.014 (0.045)
  Cluster 2: number analyzed (Participants) | 36
  Cluster 2 | -0.070 (0.048)
  Cluster 3: number analyzed (Participants) | 45
  Cluster 3 | -0.013 (0.046)
  Cluster 4: number analyzed (Participants) | 52
  Cluster 4 | -0.059 (0.040)
  Cluster 5: number analyzed (Participants) | 30
  Cluster 5 | 0.000 (0)
Statistical Analysis 1: Comparison: NutropinAq 10 mg/2 ml (30 IU); Analysis of the disease condition (GHD versus TS) on the IGF-I value as measured by capillary blood spot method; Test type: Other; F value = 10.73; For the effect of the disease condition on the IGF-I levels; F value = 10.73 and the significance probability value, PR>F = 0.0012
Statistical Analysis 2: Comparison: NutropinAq 10 mg/2 ml (30 IU); Analysis of the country cluster on the IGF-I value as measured by capillary blood spot method; Test type: Other; F value = 2.20; For the effect of the country cluster on the IGF-I levels; F value = 2.20 and the significance probability value, PR>F = 0.0701

5. Secondary Outcome: Multivariate Linear Regression Analyses to Assess Factors Affecting the Variability of IGF-I Levels: Categorised by Time of Year, Calculated Age at Enrolment and Disease Condition
Description: A multivariate linear regression analysis of factors on WCV using a stepwise forward-backward elimination was used to determine the effect of individual factors on IGF-I values as measured using the capillary blood spot method (p=0.15 for a variable to enter and remain in the model). The WCV was computed from the series of 6 measurements (2 samplings in each of Weeks 21, 22 and 23). The influence of the time of the year (1st, 2nd, 3rd and 4th quarters), calculated age at enrolment and disease condition on the IGF-I value were assessed.
  Parameter estimates from the statistical model are presented as least squares means for the categories of time of the year (1st, 2nd, 3rd and 4th quarters), calculated age at enrolment and disease condition (GHD and TS).
Time Frame: Up to Week 24
Population: The Per Protocol Population consisted of all patients in the ITT Population for whom no major protocol violations/deviations occurred. Only evaluable subjects within each of the individual subgroups are presented for each category.
Measure: Least Squares Mean (Standard Error); unit: Regression coefficient
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 175
Regression coefficient
  1st quarter | 0.118 (0.034)
  2nd quarter | 0.028 (0.033)
  3rd quarter | 0.029 (0.038)
  4th quarter | 0.000 (0)
  Calculated age at enrolment | -0.007 (0.003)
  Disease condition: GHD: number analyzed (Participants) | 106
  Disease condition: GHD | 0.051 (0.026)
  Disease condition: TS: number analyzed (Participants) | 69
  Disease condition: TS | 0.000 (0)
Statistical Analysis 1: Comparison: NutropinAq 10 mg/2 ml (30 IU); Analysis of the time of the year on the IGF-I value as measured by capillary blood spot method; Test type: Other; F value = 3.65; For the effect of the time of the year on the IGF-I levels; F value = 3.65 and the significance probability value, PR>F = 0.0139
Statistical Analysis 2: Comparison: NutropinAq 10 mg/2 ml (30 IU); Analysis of the effect of the calculated age at enrolment on the IGF-I value as measured by capillary blood spot method; Test type: Other; F value = 7.38; For the effect of the calculated age at enrolment on the IGF-I levels; F value = 7.38 and the significance probability value, PR>F = 0.0073
Statistical Analysis 3: Comparison: NutropinAq 10 mg/2 ml (30 IU); Analysis of the effect of the disease condition on the IGF-I value as measured by capillary blood spot method; Test type: Other; F value = 3.86; For the effect of the disease condition on the IGF-I levels; F value = 3.86 and the significance probability value, PR>F = 0.0511

6. Secondary Outcome: Change From Baseline at Week 24 in the IGF-I Levels as Measured by Capillary Blood Spot Method and Serum IGF-I Assay
Description: 3 simultaneous IGF-I measurements were taken at Weeks 0 (baseline), 12 and 24 by serum and capillary assay to determine the precision profile of the capillary blood spot method versus the serum IGF-I assay.
  Change from baseline at Week 24 in the IGF-I measurements by capillary blood spot method and serum assay are presented.
Time Frame: Baseline to Week 24
Population: The ITT Population consisted of all treated patients (enrolled patients who received at least one injection of treatment) and who provided any follow-up data. Evaluable subjects with data available at Week 24 are presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
ng/mL
  IGF-I Capillary blood spot method: number analyzed (Participants) | 219
  IGF-I Capillary blood spot method | 123.49 (127.40)
  Serum IGF-I assay: number analyzed (Participants) | 151
  Serum IGF-I assay | 215.41 (188.03)
Statistical Analysis 1: Comparison: NutropinAq 10 mg/2 ml (30 IU); The Bland and Altman method was used to compare the results of each of the three simultaneous random capillary and serum measurements were compared. The difference between the capillary blood spot method and the serum IGF-I measurements is presented; Test type: Other; Mean difference = -164.79, 95% CI 2-sided [-483.35 to -153.77], Standard Error of Mean 159.28

7. Secondary Outcome: Change From Baseline at Week 12 and Week 24 in Insulin-Like Growth Factor Binding Protein 3 (IGFBP3) Measurements
Description: The LWPES recommends that treatment for any indication with recombinant GH therapy in children be accompanied by regular monitoring of IGF-I and IGFBP3 concentrations. IGFBP3 binds circulating IGF-I and serum samples were taken at Visit 1 (Week 0), Visit 2 (Week 12) and Visit 3 (Week 24) in order to measure IGFBP3.
  Change from baseline (Visit 1) at Visits 2 and 3 in IGFBP3 is presented.
Time Frame: Baseline to Week 12 and Week 24
Population: The ITT Population consisted of all treated patients (enrolled patients who received at least one injection of treatment) and who provided any follow-up data. Evaluable subjects with data available at each timepoint are presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
ng/mL
  Change from baseline to Visit 2: number analyzed (Participants) | 235
  Change from baseline to Visit 2 | 1112.4 (1321.4)
  Change from baseline to Visit 3: number analyzed (Participants) | 230
  Change from baseline to Visit 3 | 1285.2 (1350.9)

8. Secondary Outcome: Change From Baseline at Week 24 in the Auxological Parameter Height
Description: The auxological parameter, height, was measured at Visit 1 (Baseline measurement), Visit 2 (Week 12) and Visit 3 (Week 24).
  Change from baseline in measured height at Visit 3 (Week 24) for the overall ITT population is presented.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
cm | 4.73 (1.69)

9. Secondary Outcome: Change From Baseline at Week 24 in the Auxological Parameter Calculated Height SDS
Description: The auxological parameter, height, was measured at Visit 1 (Baseline measurement), Visit 2 (Week 12) and Visit 3 (Week 24). The French growth charts were used for the calculation of SDS parameters: the charts provide for each age range and sex a mean parameter and SD value, from which the SDS parameter can be derived assuming a normal distribution. For example: Height SDS = (height - reference mean height (age, sex)) / reference SD (age, sex). The SDS indicates the number of standard deviations away from the mean. A SDS of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. A positive change in SDS indicates an improvement in growth, therefore, a favorable outcome.
  Change from baseline in the calculated height SDS at Visit 3 (Week 24) for the overall ITT population is presented.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD Score
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
SD Score | 0.45 (0.37)

10. Secondary Outcome: Change From Baseline at Week 24 in the Auxological Parameter Weight
Description: The auxological parameter, weight, was measured at Visit 1 (Baseline measurement), Visit 2 (Week 12) and Visit 3 (Week 24).
  Change from baseline in measured weight at Visit 3 (Week 24) for the overall ITT population is presented.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
kg | 2.01 (1.87)

11. Secondary Outcome: Change From Baseline at Week 24 in the Auxological Parameter Calculated Weight SDS
Description: The auxological parameter, weight, was measured at Visit 1 (Baseline measurement), Visit 2 (Week 12) and Visit 3 (Week 24). The French growth charts were used for the calculation of SDS parameters: the charts provide for each age range and sex a mean parameter and SD value, from which the SDS parameter can be derived assuming a normal distribution. For example: Weight SDS = (weight - reference mean weight (age, sex)) / reference SD (age, sex). The SDS indicates the number of standard deviations away from the mean. A SDS of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. A positive change in SDS indicates an improvement in weight, therefore, a favorable outcome.
  Change from baseline in the calculated weight SDS at Visit 3 (Week 24) for the overall ITT population is presented.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD Score
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
SD Score | 0.20 (0.56)

12. Secondary Outcome: Change From Baseline at Week 24 in the Auxological Parameter Annualised Growth Velocity
Description: The auxological parameter, annualised growth velocity, was measured at Visit 1 (Baseline measurement), Visit 2 (Week 12) and Visit 3 (Week 24).
  Change from baseline in the measured annualised growth velocity at Visit 3 (Week 24) for the overall ITT population is presented.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
cm/year | 5.20 (4.72)

13. Secondary Outcome: Change From Baseline at Week 24 in the Auxological Parameter Annualised Growth Velocity SDS
Description: The auxological parameter, annualised growth velocity, was measured at Visit 1 (Baseline measurement), Visit 2 (Week 12) and Visit 3 (Week 24). The French growth charts were used for the calculation of SDS parameters: the charts provide for each age range and sex a mean parameter and SD value, from which the SDS parameter can be derived assuming a normal distribution. For example: Annualised GV SDS = (annualised GV - reference mean annualised GV (age, sex)) / reference SD (age, sex). The SDS indicates the number of standard deviations away from the mean. A SDS of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. A positive change in SDS indicates an improvement in growth velocity, therefore, a favorable outcome.
  Change from baseline in the annualised growth velocity SDS at Visit 3 (Week 24) for the overall ITT population is presented.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD Score
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
SD Score | 5.10 (4.80)

14. Secondary Outcome: Percentage of Patients Rating the Overall Handling of the Administration Device, NutropinAq Pen, to Assess the Acceptability and Tolerance of NutropinAq and Its Pen
Description: The acceptability was evaluated by a questionnaire at Month 5. The users (parents and/or child) of NutropinAq pen and compliance aid booklet were asked to describe and rate the pen, cartridge, compliance aid booklet and their ease of use.
  The percentage of patients responding to each category for the assessment of the overall handling of the NutropinAq pen are presented. The categories are: Very easy, Easy, Moderately difficult, Difficult, Very difficult and Missing.
Time Frame: At Month 5
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 244
Percentage of patients
  Very easy | 39.8
  Easy | 52.5
  Moderately difficult | 3.3
  Difficult | 0
  Very difficult | 0.4
  Missing | 4.1

15. Secondary Outcome: Posology of NutropinAq at Baseline (Visit 1) Summarised as Mean Dose
Description: It was intended that the posology (mg/kg/day) of NutropinAq would remain constant throughout the study. The mean posology adopted at Visit 1 is presented.
Time Frame: Visit 1 (Baseline)
Population: The Safety Population consisted of all patients who received at least one injection of treatment.
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 248
mg/kg/day | 0.0382 (0.0092)

16. Secondary Outcome: Extent of Exposure to NutropinAq Throughout the Study
Description: The extent of treatment exposure throughout the study is presented as the mean number of daily injections performed.
Time Frame: Up to Week 24
Population: The Safety Population consisted of all patients who received at least one injection of treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
Number analyzed (Participants) | 248
days | 159.7 (35.8)

ADVERSE EVENTS:
Time Frame: From baseline (Week 0) up to Week 24.
Description: Treatment emergent adverse events are presented for the Safety Population which consisted of all patients who received at least 1 injection of treatment.
Arm/Group | NutropinAq 10 mg/2 ml (30 IU)
All-Cause Mortality (participants affected / at risk) | 0/248
Serious Adverse Events (participants affected / at risk) | 6/248
Other Adverse Events (participants affected / at risk) | 81/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NutropinAq 10 mg/2 ml (30 IU) (N=248)
Bronchopneumonia (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Retinitis Pigmentosa (Congenital, familial and genetic disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NutropinAq 10 mg/2 ml (30 IU) (N=248)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Auricular swelling (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Thyroiditis acute (Endocrine disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5)
Aptyalism (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (8)
Asthenia (General disorders) | 2 (3)
Face oedema (General disorders) | 1 (1)
Feeling cold (General disorders) | 1 (1)
Hyperthermia (General disorders) | 1 (1)
Injection site bruising (General disorders) | 2 (2)
Injection site oedema (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 9 (10)
Acute sinusitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchitis acute (Infections and infestations) | 3 (3)
Bronchopneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (2)
Enterovirus infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (4)
Lower respiratory tract infection (Infections and infestations) | 2 (3)
Nasopharyngitis (Infections and infestations) | 3 (3)
Otitis media (Infections and infestations) | 5 (6)
Rhinitis (Infections and infestations) | 6 (6)
Scarlet fever (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2)
Tonsillitis bacterial (Infections and infestations) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (10)
Viral infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 2 (2)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Insulin-like Growth Factor increased (Investigations) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 14 (27)
Migraine (Nervous system disorders) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1)
Wound haemorrhage (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes